CLINICAL TRIAL: NCT03315026
Title: Phase II Study of Interleukin 6 Blockade With Siltuximab to Decrease Symptom Burden in Patients Age 60-75 Undergoing Autologous Stem Cell Transplantation for Multiple Myeloma and AL Amyloidosis
Brief Title: Siltuximab to Decrease Symptom Burden After Autologous Stem Cell Transplantation for Patients With Multiple Myeloma and AL Amyloidosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-365
Record Dates: First submitted 2017-10-13; First posted 2017-10-19 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; AL Amyloidosis
Keywords: Siltuximab; Autologous Stem Cell Transplantation (AST); 17-365
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis | interventions — siltuximab

STUDY DESIGN:
Intervention Model Description: This is a phase II study investigating the symptomatic and cytokine response to an anti-IL-6 chimeric monoclonal antibody (siltuximab) during the acute phase of autologous stem cell transplantation (ASCT) in older individuals with multiple myeloma (MM) and systemic AL amyloidosis (AL).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Siltuximab (Experimental): Siltuximab 11mg/kg will be administered seven days before and 21 days after autologous stem cell infusion (+/-2 day).
  Interventions: Drug: Siltuximab; Behavioral: The M.D. Anderson Symptom Inventory (MDASI)

INTERVENTIONS:
Drug: Siltuximab — Siltuximab at 11mg/kg will be administered as a 1-hour infusion on day -7 and day +21 (+/-2) after stem cell infusion.
Behavioral: The M.D. Anderson Symptom Inventory (MDASI) — assessments will be conducted at baseline (day -10 +/-3), day -2 (+/-1), , day +7 (+/-1 ), and day 30 (+/-3).

SUMMARY:
Autologous stem cell transplant is beneficial to patients who are diagnosed with multiple myeloma or systemic amyloidosis. However, undesired symptoms such as weakness, fatigue, nausea, pain and sleep disturbance after transplant can contribute to complications and increase the how long the patient is in the hospital, especially in patients age 60-75. Research has shown that the development and the intensity of these symptoms are closely associated with an increase in a protein called a cytokine which is involved in the inflammatory response in the human body. One of the cytokines is called Interleukin-6 or IL-6.Therefore, this study will investigate if blocking IL-6 with an agent called siltuximab, administered before and after transplant, will decrease the symptom burden after transplant to improve quality of life and recovery in the immediate post-transplant period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-confirmed symptomatic multiple myeloma or AL amyloidosis undergoing autologous HCT with melphalan 140 or 200 mg/m2
* Age 60 through 75 years
* Have at least 3 million x 10e6 CD34+ cells/kg to be infused
* Diffusion capacity >45% (adjusted for hemoglobin) as predicted by pulmonary function testing.
* KPS performance status ≥ 60% or ECOG Performance Status score of 0-2
* Clinical laboratory values meeting the following criteria within 4 weeks before enrollment:

  * LVEF >45% by MUGA or rest ECHO
  * Diffusion capacity >45% (adjusted for hemoglobin) as predicted pulmonary function testing
  * Platelet count ≥ 20 x 10^9/L
  * ALT and AST ≤ 2.5 x ULN
  * Total bilirubin ≤ 2.5 x ULN; except if the elevation is due to Gilbert's syndrome
  * Calculated creatinine clearance > 40 mL/min
* Before enrollment, all women are expected to be not of childbearing potential as they will be age 60-75>:

  * Not of childbearing potential: postmenopausal (>45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level >40 IU/mL); permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy); or otherwise be incapable of pregnancy
  * Of childbearing potential and practicing (during the study and for 3 months after receiving the last dose of study agent) a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: eg, established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; male partner sterilization (the vasectomized partner should be the sole partner for that subject); true abstinence (when this is in line with the preferred and usual lifestyle of the subject)
  * A woman of childbearing potential must have a negative serum (β-human chorionic gonadotropin [β-hCG]) pregnancy test at screening
  * During the study and for 3 months after receiving the last dose of study agent, a woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction
  * Note: If the childbearing potential changes after start of the study (eg, woman who is not heterosexually active becomes active) a woman must begin a highly effective method of birth control, as described above.
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control eg, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Prior exposure to agents targeting IL-6 or the IL-6 receptor
* Other malignancy within the past 2 years, except for the following if treated and not active: basal cell or nonmetastatic squamous cell carcinoma of the skin, cervical carcinoma in situ or International Federation of Gynecology and Obstetrics (FIGO) Stage 1 carcinoma of the cervix
* Concurrent medical condition or disease (eg, autoimmune disease, active systemic Infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in the study
* Vaccination with live attenuated vaccines within 4 weeks of first study agent administration
* Clinically significant infection, including known HIV or hepatitis C infection, or known hepatitis B (Hep B) surface antigen positivity. Patients with Hep B Core positivity can be enrolled if the Hep B PCR is negative, and they are on antiviral suppression.
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 14 days or 5 half lives before enrollment or is currently enrolled in the treatment stage of an investigational study
* Had hospitalization for infection or major surgery (eg, requiring general anesthesia) within 2 weeks before enrollment or have not fully recovered from surgery. Note: subjects with surgical procedures conducted under local anesthesia may participate
* A woman who is pregnant or breast-feeding, or a woman who is planning to become pregnant or a man who plans to father a child while enrolled in this study or within 3 months after the last dose of study agent.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
number of patients with improved symptoms | 30 days post ASCT
  as assessed by the MD Anderson symptom inventory Multiple Myeloma Module (MDASI-MM)

CONTACTS AND LOCATIONS:
Overall Officials: Gunjan Shah, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm